CLINICAL TRIAL: NCT02790476
Title: Use of Behavioral Insights to Encourage Judicious Prescribing of Opioids
Brief Title: Behavioral Insights to Encourage Judicious Prescribing of Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jason Doctor, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHCF-16-00053
Record Dates: First submitted 2016-05-27; First posted 2016-06-06 (Estimated); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Substance-Related Disorders
Keywords: Safe; Prescribing; Opioids
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letter intervention (Experimental): The intervention arm will involve letters sent to prescribers in San Diego County.
  Interventions: Other: Letters
- Control (No Intervention): The control group will involve prescribers not receiving letters

INTERVENTIONS:
Other: Letters — The letters will be factual and nonjudgmental, signed by the County Medical Examiner, and would state that a patient they had treated with controlled substances died of an opioid poisoning. The letter will encourage judicious prescribing, and will provide information developed by an advisory group: how to identify and taper unsafe regimens (high dose, polypharmacy, or use of multiple prescribers); how to identify addiction and compassionately refer patients for medication-assisted treatment; and recommendations to avoid bad outcomes (e.g. "do not fire your patient for signs of addiction.") The letter would also encourage use of the CURES system before prescribing, as well as co-prescribing of naloxone.
  Arms: Letter intervention

SUMMARY:
In collaboration with the San Diego Medical Examiner's Office and the State of California's controlled Substance Utilization Review and Evaluation System (CURES), the investigators propose to review opioid poisonings over the past 12 months and will send letters to prescribers in California when at least one of the provider's prescription(s) was filled by a patient who died of an opioid poisoning in San Diego County. The letters will be non-judgmental and factual, explaining that a patient of the provider who was being treated with prescription narcotics died of an opioid poisoning. The letter will also encourage judicious prescribing including use of the CURES system before prescribing. The investigators will evaluate physician prescribing practices over 24 months 12 months pre- and 12 months post-letter using data from the CURES database. The investigators' hypothesis is that letters will make the risk of opioids more cognitively available and that physicians will respond by prescribing opioids more carefully. This will result in fewer deaths due to misuse and more frequent use of the CURES system.

ELIGIBILITY:
The investigators will not be enrolling subjects. This is an evaluation of a public health intervention involving sending prescriber's factual and nonjudgmental letters, signed by the County Medical Examiner, that would state that a patient the provider had treated with controlled substances died of an opioid poisoning.

Inclusion Criteria:

* Prescribers in California for whom at least one of their prescription(s) was filled by a patient who died of an opioid poisoning in San Diego County

Exclusion Criteria:

* Prescriber is licensed outside the State of California and does not hold a California license, but the prescription was filled in California
* The prescriber does not have a CURES report on record
* The prescriber has issued only one opioid prescription in the last 12 months since the time of the deceased death (and the prescription was to the deceased)
* Prescribers with unknown Drug Enforcement Agency number

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-05-27 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- San Diego County Medical Examiner's Office, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Letter Intervention | Control
Started | 404 | 447
Completed | 386 | 425
Not Completed | 18 | 22

BASELINE CHARACTERISTICS:
Population: We removed prescribers with missing data or lack of prescriptions during the study period, resulting in an analysis population of 811 prescribers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Letter Intervention | Control | Total
Number analyzed (Participants) | 386 | 425 | 811
Age, Categorical [Count of Participants; unit: Participants] — Population: We did not collect data on age of prescribers.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We did not collect data on biological sex from prescribers.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 386 | 425 | 811

OUTCOME MEASURES:

1. Primary Outcome: Average Change Over Time in Dispensed Narcotics
Description: The hypothesis is that the average change over time in dispensed narcotic represented as monthly morphine milligram equivalent (MME) dose will be larger for prescribers receiving the letter intervention, compared to the average change over time for the control prescribers not receiving the letter intervention.
Time Frame: 12 months
Population: Clinicians and allied health professionals with scheduled drug prescribing privileges in California who prescribed a schedule II, III, or IV drug to a person who died as a result of a schedule II, III, or IV accidental overdose between the period of 1 July 2015 and 30 June 2016 in San Diego County.
Measure: Mean (95% Confidence Interval); unit: Morphine milligram equivalents
Arm/Group | Letter Intervention | Control
Number analyzed (Participants) | 386 | 425
Morphine milligram equivalents
  Adjusted per-prescriber mean weekly morphine milligram equivalents (MMEs); Pre intervention | 347.65 [339.27 to 356.03] | 350.09 [341.77 to 358.40]
  Adjusted per-prescriber mean weekly MMEs; 1-3 months Post intervention | 288.36 [281.61 to 295.11] | 318.60 [311.03 to 326.17]
  Adjusted per-prescriber mean weekly MMEs; 4-12 months Post intervention | 167.83 [163.91 to 171.74] | 182.67 [178.46 to 186.88]
Statistical Analysis 1: Comparison: Letter Intervention; 1-3 months post intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -27.80, 95% CI 2-sided [-38.20 to -17.63] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (288.36-347.65 = -59.29) and control (318.60-350.09 = -31.49) arms, resulting in a difference of -27.80
Statistical Analysis 2: Comparison: Letter Intervention; Test type: Superiority; p < 0.01, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -12.42, 95% CI 2-sided [-18.40 to -6.55] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (167.83-347.65 = -179.83) and control (182.67-350.09 = -167.41) arms, resulting in a difference of -12.42

2. Primary Outcome: Number of Opioid Prescriptions for > 90 Morphine Milligram Equivalent (MME) and ≥ 50 MME
Description: The hypothesis is that there will be fewer opioid prescriptions both at a dose > 90 morphine milligram equivalent (MME) and at a dose ≥ 50 MME among prescribers receiving the letter intervention, compared to control prescribers not receiving the letter intervention.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Number of prescriptions
Arm/Group | Letter Intervention | Control
Number analyzed (Participants) | 386 | 425
Number of prescriptions
  Number of => 50 MME Prescriptions Pre intervention | 3.74 [3.57 to 3.91] | 4.59 [4.41 to 4.76]
  Number of => 50 MME Prescriptions 1-3 months Post intervention | 3.45 [3.08 to 3.82] | 3.95 [3.59 to 4.30]
  Number of => 50 MME Prescriptions 4-12 months Post-intervention | 3.00 [2.79 to 3.21] | 3.15 [2.95 to 3.35]
  Number of > 90 MME Prescriptions Pre intervention | 2.14 [2.02 to 2.27] | 2.55 [2.44 to 2.67]
  Number of > 90 MME Prescriptions 1-3 Post intervention | 2.00 [1.76 to 2.25] | 2.20 [1.96 to 2.44]
  Number of > 90 MME Prescriptions 4-12 months Post intervention | 1.71 [1.57 to 1.85] | 1.74 [1.61 to 1.87]
Statistical Analysis 1: Comparison: Letter Intervention; Change in mean number of => 50 MME prescriptions pre- to 1-3 months post-intervention; Test type: Superiority; p = 0.224, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.92 to 0.22] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (3.45-3.74 = -0.29) and control (3.45-4.59= -0.64) arms, resulting in a difference of -0.35
Statistical Analysis 2: Comparison: Letter Intervention; Change in mean number of => 50 MME prescriptions pre- to 4-12 months post-intervention; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.08 to -0.33] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (3.00-3.74 = -0.74) and control (3.15-4.59= -1.44) arms, resulting in a difference of -0.70
Statistical Analysis 3: Comparison: Letter Intervention; Change in mean number of > 90 MME prescriptions pre- to 1-3 months post-intervention; Test type: Superiority; p = 0.279, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.59 to 0.17] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (2.00-2.14 = -0.14) and control (2.20-2.55= -0.35) arms, resulting in a difference of -0.21
Statistical Analysis 4: Comparison: Letter Intervention; Change in mean number of > 90 MME prescriptions pre- to 4-12 months post-intervention; Test type: Superiority; p < 0.01, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.63 to -0.12] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (1.71-2.14 = -0.43) and control (1.74-2.55= -0.81) arms, resulting in a difference of -0.38

3. Primary Outcome: Number of Opioid and Benzodiazepine Co-prescriptions
Description: The hypothesis is that there will be fewer opioid and benzodiazepine co-prescriptions for prescribers receiving the letter intervention, compared to control prescribers not receiving the letter intervention.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Adjusted mean number of co-prescriptions
Arm/Group | Letter Intervention | Control
Number analyzed (Participants) | 352 | 390
Adjusted mean number of co-prescriptions
  Pre intervention | 12.2 [9.8 to 14.6] | 13.6 [11.0 to 16.1]
  Post intervention | 13.4 [12.3 to 14.4] | 16.7 [15.5 to 17.9]
Statistical Analysis 1: Comparison: Letter Intervention; Test type: Superiority; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Pre-intervention values were trimmed at 95% with bootstrapped means and confidence intervals; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.2 to -0.1] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean DME in the letter (72.3-76 = -3.7) and control (82-82.9 = -0.9) arms, resulting in a difference of -1.6

4. Secondary Outcome: Frequency of CURES Use
Description: The hypothesis is that there will be more frequent use of CURES among prescribers receiving the letter intervention, compared to control prescribers not receiving the letter intervention.
Time Frame: 12 months
Population: We were unable to access information on frequency of CURES use and could not conduct the proposed analysis.
Arm/Group | Letter Intervention | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of "New Start" Prescriptions
Description: The hypothesis is that there will be fewer prescriptions for opioid naïve patients by prescribers receiving the letter intervention, compared to control prescribers not receiving the letter intervention.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: patients with new opioid prescriptions
Arm/Group | Letter Intervention | Control
Number analyzed (Participants) | 386 | 425
patients with new opioid prescriptions
  Pre intervention | 3.72 [3.64 to 3.80] | 3.51 [3.44 to 3.59]
  1-3 months post intervention | 2.44 [2.27 to 2.61] | 2.26 [2.10 to 2.43]
  4-12 months post intervention | 2.08 [1.99 to 2.18] | 1.84 [1.76 to 1.93]
Statistical Analysis 1: Comparison: Letter Intervention; Change in mean number of new patients pre- to 1-3 months post-intervention; Test type: Superiority; p = 0.823, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.23 to 0.29] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (2.44-3.72 = -1.28) and control (2.26-3.51= -1.25) arms, resulting in a difference of 0.03
Statistical Analysis 2: Comparison: Letter Intervention; Change in mean number of new patients pre- to 4-12 months post-intervention; Test type: Superiority; p = 0.692, Mixed Models Analysis — The threshold for statistical significance is p=0.05; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.20 to 0.14] — This measure is a difference-in-difference, calculated by subtracting the pre- and post-intervention difference in mean MME in the letter (2.08-3.72 = -1.64) and control (1.84-3.51= -1.67) arms, resulting in a difference of -0.03

ADVERSE EVENTS:
Time Frame: 12 months following letter notification (January 28, 2017-January 27, 2018)
Arm/Group | Letter Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/386 | 0/425
Serious Adverse Events (participants affected / at risk) | 0/386 | 0/425
Other Adverse Events (participants affected / at risk) | 0/386 | 0/425

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT02790476/Prot_SAP_000.pdf